CLINICAL TRIAL: NCT04592159
Title: A Randomized, Double-blind, Parallel-group Study of the Safety and Efficacy of Nabiximols Oromucosal Spray Versus Placebo in Patients With Post-traumatic Stress Disorder
Brief Title: Study of the Safety and Efficacy of Nabiximols Oromucosal Spray Versus Placebo in Patients With Post-traumatic Stress Disorder
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The decision to suspend this study was based upon evaluation of pandemic-related challenges impacting both clinical trial sites and potential participants. This suspension was initiated prior to site activation and participant recruitment.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GWPD19177; 2020-000527-39 (EudraCT Number)
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Nabiximols; Selective serotonin reuptake inhibitor; Serotonin-norepinephrine reuptake inhibitor
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nabiximols (Experimental): Nabiximols is a complex botanical medicine formulated from extracts of the cannabis plant that contains the principal cannabinoids delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD) and also contains minor constituents, including other cannabinoid and non-cannabinoid plant components, such as terpenes, sterols, and triglycerides.Each spray delivers 100 microliters (μL) of nabiximols.
  Interventions: Drug: Nabiximols
- Placebo (Placebo Comparator): Placebo to match nabiximols will be presented as an oromucosal spray containing the excipients ethanol and propylene glycol (50% v/v) with colorings and flavored with peppermint oil (0.05% v/v). Each spray will deliver 100 μL containing no active ingredients. Placebo will be self-administered by participants as an oromucosal spray in the morning and evening, up to a maximum of 12 sprays per day for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nabiximols — oromucosal spray
  Other Names: GW-1000-02; Sativex
  Arms: Nabiximols
Drug: Placebo — oromucosal spray
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the efficacy of nabiximols for the treatment of symptoms of post-traumatic stress disorder (PTSD) in participants receiving selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) pharmacotherapy.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled, parallel-group trial includes a screening period of up to 28 days, an 8-week treatment period (comprising a 2-week titration phase and a 6-week maintenance phase), and a 2-week follow-up period.

At screening (Visit 1), all participants will receive instructions on how to complete a writing exercise (Exposure Writing Exercise) related to their traumatic experience. Prior to the baseline visit (Visit 2), participants must complete an approximate 30-minute writing exercise outside of the trial site and should have re-read the write up at least once to be eligible for enrollment.

Throughout the screening and treatment periods, the dose of SSRI/SNRI used as background therapy, if any, should remain unchanged. On Day 1, eligible participants will be randomly assigned to either nabiximols or placebo in a 1:1 ratio.

Participants will be advised to titrate the investigational medicinal product (IMP), beginning with 1 spray/day, to an optimized dose that relieves their most bothersome symptom of PTSD or to a maximum of 12 sprays/day over the first 14 days of treatment. Participants should continue at the same dose level achieved at the end of the titration phase ±1 spray divided into a morning dose and an evening dose for the remainder of the treatment period.

Health-related quality of life, safety, and tolerability will be evaluated during the treatment period.

Participants who complete the trial will participate for a total of approximately 14 weeks (99 days), including the 28-day Screening period.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders, Volume 5 (DSM-5) criteria for post-traumatic stress disorder (PTSD), confirmed on the basis of the Mini International Neuropsychiatric Interview (MINI)
* If currently taking a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for the treatment of PTSD, SSRI/SNRI doses should be consistent with approved labelling and have been stable for at least 6 weeks prior to Visit 1 with no more than 1 SSRI/SNRI.
* If not currently taking a SSRI or SNRI, should not have received treatment with either a SSRI or SNRI for at least 6 weeks prior to Visit 1 and is not planning to start additional pharmacotherapy during the study
* Exhibits significant PTSD symptoms and associated impairment (as reflected by Clinician Administered PTSD Scale [CAPS-5] ≥ 27 and Clinical Global Impressions Severity [CGI-S] ≥ 4 at Visit 1), which should have persisted over a period of at least 3 months prior to Visit 1
* Willing to allow the responsible authorities to be notified of participation in the trial, if mandated by local law
* Willing to allow his or her primary care practitioner (if they have one) and consultant (if they have one) to be notified of participation in the trial, if the primary care practitioner/consultant is different to the investigator

Exclusion Criteria:

* Is at risk of suicide as evidenced by a history of suicide attempt(s) in the 2 years prior to Visit 1 or answering yes on item 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) in the month prior to Visit 1
* Is currently involved in any legal action that relates to the diagnosis of PTSD or the traumatic events that gave rise to the disease
* Has cognitive impairment that in the opinion of the investigator may interfere with participation in the study or ability to complete assessments or report treatment effects
* Has any history of psychosis (including schizophrenia, schizophreniform disorder, schizoaffective disorder, or substance-induced psychosis), or bipolar disorder based on an assessment using the MINI.
* Participants who have an index trauma before age 18 and no other traumatic experiences which could relate/identify as being part of their PTSD
* Has taken cannabis or a cannabis derived product for medicinal or recreational purposes at any time in the past and developed significant adverse experiences related to cannabis use per history and investigator judgment
* Has severe depressive symptoms as per the investigator's judgment or a score ≥ 20 on the Patient Health Questionnaire-9 (PHQ-9) at Visit 1
* Has a history of any degree of DSM-5 cannabis or other substance use disorder, or moderate to severe alcohol use disorder within 6 months prior to Visit 1. Participants with Nicotine Use Disorder are allowed to enroll.
* Has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal product
* Has recently taken nabiximols, cannabis, or a cannabis-derived product for medicinal or recreational purposes as reflected by a positive Δ9-tetrahydrocannabinol (THC) urine test at Visit 1
* Currently taking 1 of a number of specified psychotropic medications, where there is a potential for pharmacodynamic interactions. Participants taking any medication with psychoactive properties not currently on the list of prohibitive medications may be considered for enrollment only after consultation with a GW medical representative.
* Has experienced myocardial infarction or clinically significant cardiac dysfunction within the 12 months prior to Visit 1 or has a cardiac disorder that, in the opinion of the investigator, would put the participant at risk of a clinically significant arrhythmia or myocardial infarction
* Positive serology panel (including hepatitis B surface antigen [HBsAg] and hepatitis C virus [HCV] antibody)
* Positive human immunodeficiency virus (HIV) antibody/p24 antigen screens
* Has a diastolic blood pressure of < 50 millimeters of mercury (mmHg) or > 105 mmHg or systolic blood pressure < 90 mmHg or > 150 mmHg (when measured in a sitting position at rest for 5 minutes) or a postural drop in the systolic blood pressure of > 20 mmHg at Visit 1
* Has clinically significant impaired renal function at Visit 1, as evidenced by an estimated creatinine clearance lower than 50 milliliters per minute (mL/min)
* Has serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) at Visit 1
* Male and fertile (i.e., after puberty unless permanently sterile by bilateral orchiectomy) unless willing to ensure that he uses male contraception (condom or vasectomy) or remains sexually abstinent during the trial and for 3 months thereafter
* Female and of childbearing potential (i.e., following menarche and until becoming postmenopausal for ≥ 12 consecutive months unless permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) unless willing to ensure that she uses a highly effective method of birth control (e.g., intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomized partner, or sexual abstinence) during the trial and for 3 months thereafter. Participants using combined hormonal methods or a progestogen-only pill or injection or implant should use an additional barrier method such as a male condom or diaphragm during the trial and for 3 months thereafter.
* Female and pregnant (positive pregnancy test at Visit 1), lactating, or planning pregnancy during the course of the trial or within 3 months thereafter
* Has participated in an interventional or non-interventional clinical trial within the 30 days prior to Visit 1
* Has donated blood during the 3 months prior to Visit 1 and is unwilling to abstain from donation of blood during the trial
* Has been previously randomized into this trial
* Any abnormalities identified following a physical examination, clinical laboratory, serology, or other applicable screen procedures that, in the opinion of the investigator, would jeopardize the safety of the participant or the conduct of the study if they took part in the trial
* Participants who are currently participating in a trauma-focused psychotherapy are ineligible to participate in the trial. Participants who are participating in other forms of psychotherapy (or none at all) must agree to continue (or not start) therapy during the trial.

Additional exclusion criterion at Visit 2 (Day 1, pre-randomization):

* Exhibited a CAPS-5 score < 27 at Visit 2, or a reduction in CAPS-5 score of ≥ 30% at Visit 2 relative to Visit 1
* Did not complete the writing exercise during the screening period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinician Administered Post-Traumatic Stress Disorder (PTSD) Scale (Clinician Administered PTSD Scale [CAPS-5]) Score over 8 Weeks | Baseline; Week 8

SECONDARY OUTCOMES:
Number of Participants Exhibiting Improvements Rated as Much or Very Much Improved on the Clinical Global Impressions Improvement (CGI-I) Scale at the End of Treatment (over 8 Weeks) | from Baseline up to Week 8
Change from Baseline in the Self-Reported PTSD Checklist for the Diagnostic and Statistical Manual of Mental Disorders, Volume 5 (DSM-5) (PCL-5) Score over 8 Weeks | Baseline; Week 8
Number of Participants with any Treatment-Emergent Adverse Event | up to Week 8
Number of Participants with the Indicated Change from Baseline in Clinical Laboratory Test Values | Baseline; Week 8
Change from Baseline in Systolic Blood Pressure | Baseline; Week 8
Change from Baseline in Diastolic Blood Pressure | Baseline; Week 8
Change from Baseline in Pulse Rate | Baseline; Week 8
Number of Participants with Clinically Significant 12-Lead Electrocardiogram (ECG) Parameter Values | from Baseline up to 8 weeks
Change from Baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS) Score | Baseline; Week 8

IPD SHARING:
Plan to Share IPD: No